CLINICAL TRIAL: NCT00964769
Title: A Study of Evaluation Indexes for Antibody Production in Sera After Immunization
Brief Title: Study of Evaluation Indexes for Antibody Production in Sera After Immunization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Kyung-Hyo Kim, Ewha Womans Univrsity Hospital
Model: Parallel | Masking: None
Other Study IDs: EU-KF-05092341; 05092KFDA341
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Aged
Keywords: Pneumococcal Vaccine; Aged
MeSH Terms: interventions — Pneumococcal Vaccines; 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pneumococcal polysaccharide vaccine (Experimental): The immunogenic response to the pneumococcal polysaccharide vaccine was compared between children, adults and elderly.
  Interventions: Biological: pneumococcal polysaccharide vaccine

INTERVENTIONS:
Biological: pneumococcal polysaccharide vaccine — single intramuscular injection of 0.5 ml Pneumo23® (Sanofi-Aventis, Lyon France)
  Other Names: Pneumo23®

SUMMARY:
The aim of this study is to evaluate analytical methods such as ELISA and OPKA that measure the activity of vaccine-induced pneumococcal antibodies. After validation of ELISA and OPKA, pneumococcal antibodies were measured by ELISA and OPKA in paired samples before and after immunization (pneumococcal PS vaccine) in children, adults and elderly.

DETAILED DESCRIPTION:
To evaluate the immune response to the pneumococcal polysaccharide vaccine in the elderly, samples from children, young adults and elderly were obtained before and one month after vaccination. The quantitative and qualitative response to the vaccine were measured by the ELISA and opsonophagocytic killing assay for eight vaccine type serotypes (4, 6B, 9V, 14, 18C, 19A, 19F, 23F) and one vaccine-related serotype (6A).

ELIGIBILITY:
Inclusion Criteria:

* elderly subjects over the age 65 years who had not received pneumococcal vaccination
* adult subjects under the age of 45 years (healthy volunteers with no previous history of pneumococcal vaccination)
* children subjects over the age of 2 years with no previous history of pneumococcal vaccination

Exclusion Criteria:

* immunocompromised, asplenia, cancer, liver or renal failure, and history of hypersensitivity to vaccine

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-04; Primary Completion 2005-05 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the immune response to the pneumococcal polysaccharide vaccine in children, young adults and elderly. | 1 month after vaccination

SECONDARY OUTCOMES:
Evaluate the immune response to the pneumococcal polysaccharide vaccine with two methods (ELISA and Opsonophagocytic Killing Assay) | 1 month after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Hyo Kim, Doctor, Principal Investigator — Ewha Womans University Dongdaemun Hospital
Locations (1):
- Ewha Womans University Dongdaemun Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Lee H, Nahm MH, Kim KH. The effect of age on the response to the pneumococcal polysaccharide vaccine. BMC Infect Dis. 2010 Mar 10;10:60. doi: 10.1186/1471-2334-10-60. PMID 20219110